CLINICAL TRIAL: NCT03395652
Title: Maternal Physical Activity and Pregnancy Outcome
Status: Withdrawn | Type: Observational
Why Stopped: technical problems
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Principal Investigator, marija simic, Principal Investigator, Karolinska Institutet
Other Study IDs: Karolinskal
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Complications
Keywords: pregnancy, physical activity, fetal growth
MeSH Terms: conditions — Pregnancy Complications; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the impact of maternal physical activity during pregnancy on pregnancy outcome. Primary, fetal growth during pregnancy abd birth weight will be examined.

DETAILED DESCRIPTION:
During this study, the information on maternal physical activity will be collected and the impact on delivery and pregnancy complications as well as on neonatal complications will be evaluated. From the first visit at maternal care center, the information on socioeconomical and maternal characteristics will be collected. During pregnancy, fetal growth will be estimated by ultrasound. Physical activity will be measured using free app for measuring steps that mothers make during pregnancy. Using logistic regression, the impact of physical activity on pregnancy outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Healthy women with singleton pregnancies

-

Exclusion Criteria:

* Twins pregnancies. Mothers with preexisting conditions. Malformations.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mothers included in the study live in Belgrade, Serbia and are pregnant during 2018. They are asked to participate in the study at first ultrasound examination at week 12-14.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Fetal growth | birth weight at birth
  Large for gestational age (LGA) small for gestational age (SGA)

SECONDARY OUTCOMES:
Pregnancy complications | during pregnancy ( 9 months from start)
  preeclampsia, diabetes, weight gain.